CLINICAL TRIAL: NCT03195972
Title: Observational Study to Assess Adherence of Oral Anticancer Therapies
Brief Title: Observational Study to Assess Adherence Oral Anticancer Therapies
Acronym: ObservAG
Status: Completed | Type: Observational
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Other Study IDs: ObservAG
Record Dates: First submitted 2017-06-09; First posted 2017-06-22 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Adherence, Patient
Keywords: Adherence, Patient, oncology, oral therapy
MeSH Terms: conditions — Patient Compliance; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Drug diary filling — patient will fill every day a drug diary

SUMMARY:
Oral anticancer treatments are increasingly numerous. They represent an additional alternative in the therapeutic arsenal of the clinician, and appear to satisfy patients who prefer this route of administration over intravenous treatment. The objective of oral therapies is twofold: to remove the constraints and risks associated with infusions and to allow the patient to follow his treatment at home.

However, they have significant adverse effects that may affect patients, who are sometimes at a disadvantage compared to how they are treated, and potentially lead to non-compliance with the consequences.

This study will identify the factors associated with non-adherence and determine the impact of this non-adherence in terms of treatment efficacy and tolerance.

The aim of this routine care study is to evaluate the adherence to oral anticancer therapies during 3 months.

DETAILED DESCRIPTION:
Primary objective

- To evaluate adherence to oral anti-cancer therapies at 3 months

Secondary objectives

* To evaluate the adherence to 3 months according to the age of the patients (less than 75 years versus 75 years and more)
* Evaluate compliance at 1 and 2 months
* Evaluate toxicity at 1, 2 and 3 months according to compliance according to criteria CTCAE 4.03.
* Evaluate response to treatment at 3 months based on adherence
* Evaluate the factors associated with adherence and describe the reasons for non-adherence.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* Cancer proved histologically.
* Patient receiving an initial prescription for oral anticancer therapy, excluding hormone therapy
* Illness measurable or assessable by imaging
* Patient affiliated to a social security scheme
* Patient having been informed of the study
* Non-opposition of the patient

Exclusion Criteria:

* Contraindication to oral treatment
* Patient's refusal
* Patient under tutelage, curatorship or safeguard of justice
* Psychiatric illness and / or condition of the patient compromising understanding of information or conduct of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient with cancer treated with oral therapy (targeted therapy or chemotherapy) excluding hormone therapy.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-12-23 (Actual); Primary Completion 2016-12-23 (Actual); Study Completion 2018-09-04 (Actual)

PRIMARY OUTCOMES:
Compliance with treatment | 3 months
  Treatment adherence will be assessed by the number of treatment units taken in relation to the prescribed amount. A patient will be considered as observing if he has received at least 80% of the dose initially prescribed.

SECONDARY OUTCOMES:
Toxicity | 3 months
  The toxicity of the treatment will be assessed and graded, at each medical consultation, according to the classification NCI-CTCAE V4.03, in observing and non-observing patients.
Response to treatment | 3 months
  Treatment response will be assessed according to clinical status and radiological criteria RECIST 1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- CGFL, Dijon, France

IPD SHARING:
Plan to Share IPD: No